CLINICAL TRIAL: NCT05343793
Title: Stagewise Implementation-To-Target- Medications for Addiction Treatment (SITT-MAT)
Acronym: SITT-MAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Wisconsin, Madison (Other); National Institute on Drug Abuse (NIDA) (NIH); Washington State Health Care Authority (Unknown)
Responsible Party: Principal Investigator, Mark McGovern, Professor, Stanford University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 60711; 1R01DA052975-01A1 (NIH)
Record Dates: First submitted 2022-04-06; First posted 2022-04-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Addiction, Opioid
Keywords: Implementation strategies; Medications for opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Path 1 (Experimental): Enhanced Monitoring and Feedback
  Interventions: Other: Enhanced Monitoring and Feedback (EMF)
- Path 2 (Experimental): Enhanced Monitoring and Feedback + NIATx/MAT Academy
  Interventions: Other: Enhanced Monitoring and Feedback (EMF); Other: NIATx/MAT Academy
- Path 3 (Experimental): Enhanced Monitoring and Feedback + NIATx/MAT Academy + NIATx External Facilitation
  Interventions: Other: Enhanced Monitoring and Feedback (EMF); Other: NIATx/MAT Academy; Other: NIATx-External Facilitation (NIATx-EF)
- Path 4 (Experimental): Enhanced Monitoring and Feedback + NIATx/MAT Academy + NIATx Internal Facilitation
  Interventions: Other: Enhanced Monitoring and Feedback (EMF); Other: NIATx/MAT Academy; Other: NIATx-Internal Facilitation (NIATx-IF)
- Path 5 (Experimental): Enhanced Monitoring and Feedback + NIATx/MAT Academy + NIATx Internal Facilitation + NIATx External Facilitation
  Interventions: Other: Enhanced Monitoring and Feedback (EMF); Other: NIATx/MAT Academy; Other: NIATx-Internal Facilitation (NIATx-IF); Other: NIATx-External Facilitation (NIATx-EF)

INTERVENTIONS:
Other: Enhanced Monitoring and Feedback (EMF) — Enhanced Monitoring and Feedback consists of performance data (reach, adoption, effectiveness, implementation) gathered and reported by the program on a quarterly basis. Data summaries for each program and in comparison to the entire sample, will be reflected back to participants, via dashboards, within one-month of data submission.
Other: NIATx/MAT Academy — This two-day workshop will provide participating clinics with rationale, clinical practice and program integration with MOUD (Day 1), and an overview of NIATx principles and tools (Day 2).
  Arms: Path 2; Path 3; Path 4; Path 5
Other: NIATx-Internal Facilitation (NIATx-IF) — Internal facilitators will receive training (in-person or online) on how to provide coaching within their organization. For 9-months, Internal Facilitators (IFs) will: a) support teams to harness resources toward systemic change and improvement; b) employ a range of concepts and tools to provide individualized support to teams; c) help teams to practice and hone their skills to optimize performance, and d) focus on team relationships and communications.
  Arms: Path 4; Path 5
Other: NIATx-External Facilitation (NIATx-EF) — For 9-months, organizations in the NIATx-EF study arm will work with one of 4 experienced consultant NIATx External Facilitators (EFs). The EF meets with clinic staff to plan change projects, review ongoing change efforts, discuss successes, and offer guidance on planning future change projects using PDSA cycles. The EF makes a 1-day site visit during the 1st quarter of the implementation period and leads monthly 1-hour phone calls.
  Arms: Path 3; Path 5

SUMMARY:
The purpose of this study is to expand access to medications for opioid use disorder (MOUD) in specialty addiction programs in Washington State. Sixty-four addiction treatment programs will participate in an adaptive implementation strategy trial that uses a stagewise implementation-to-target (stepped "care" type) approach whereby organizations engage in increasingly intensive implementation strategies as needed. Organizations are moved to a follow-up/sustainment arm once they have met the implementation targets described below. The design also includes an external comparator arm, which consists of 510 addiction treatment programs that are not participating in the study and will mimic as study controls.

The sequence of implementation strategies are:

1. Enhanced Monitoring and Feedback
2. NIATx/MAT Academy
3. Randomization to either NIATx Internal Facilitation or NIATx External Facilitation
4. Assignment to NIATx External Facilitation if outcome targets are not achieved in the NIATx Internal Facilitation arm

Implementation targets are:

1. Reach - At least 75% of patients with opioid use disorder (OUD) receiving MOUD for three consecutive months
2. Adoption - At least 1 integrated MOUD prescriber actively prescribing MOUD
3. Implementation - a total score ≥ 4 on the Integrating Medications for Addiction Treatment (IMAT) Index.

Contextual moderators and mediators of performance on target outcomes as a function of the implementation strategy step will be examined, as will the costs associated with participation in the sequence of implementation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Addiction treatment programs in Washington State
* Residential (detoxification or rehabilitation) or outpatient (intensive outpatient or outpatient) levels of care
* Primary care clinics, including Federally Qualified Health Centers (FQHCs) and Community Health Centers (CHCs)

Exclusion Criteria:

* Opioid treatment programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reach | Quarterly ; Months 1 to 46
  The proportion of program patients with OUD and receiving MOUD (buprenorphine, naltrexone) within the index quarter.
Adoption | Quarterly ; Months 1 to 46
  The number of integrated prescribers of buprenorphine and/or naltrexone, who are actively prescribing MOUD.
Effectiveness | Quarterly ; Months 1 to 46
  Access: The proportion of patients prescribed MOUD who start the medication within 72 hours of diagnosis. For patients requiring detoxification for naltrexone, Access will be operationalized as the proportion of patients who start the medication within 72 hours of when it is safe or indicated by a physician. Retention: The proportion of patients who are retained in continuous care for at least 6-months from the start of medication, or if in time limited care situations (e.g., residential detoxification) for the entire treatment episode.
Implementation - Integrating Medications for Addiction Treatment (IMAT) Index | Months 1,7,14,24,34,46
  The IMAT integrates MOUD guidelines, expert consensus recommendations, the OUD care cascade, and best practice information into a team-assessment benchmark measure of current and future state MOUD capability and practice. The IMAT is composed of 45 items, rated on a 1 to 5 scale from: 1- Not Integrated, to 3- Partially integrated, to 5- Fully integrated. Intermediate ratings of 2 and 4, are ratings not at either a 3 or 5 level respectively. The benchmark items address policy, practice and workforce factors, and are clustered into seven dimensions of: 1) Infrastructure; 2) Clinic culture and environment; 3) Patient identification and initiating care; 4) Care delivery and treatment response monitoring; 5) Care coordination; 6) Workforce; and, 7) Staff training and development. The IMAT Total Score is a composite rating from 1 to 5 of overall MOUD care quality. It takes between 1 to 2 hours to complete.

OTHER OUTCOMES:
Contextual determinants | Months 1,7,14,24,34,46
  Inventory of Factors Affecting Successful Implementation and Sustainment (IFASIS). The IFASIS evaluates contextual aspects at baseline and over time. This measure focuses on four dimensions (Outer Context, Inner Context, Perception of Intervention, Perception of Patient/Client Experience). tHE IFASIS is a team-assessment measure completed by key staff in MOUD implementation. In addition to individual item scores, it generates a score for each of the four dimensions and in total.
Engagement in implementation | Monthly ; Months 1 to 46
  Stages of Implementation Completion (SIC). The SIC is an 8-stage assessment tool designed to measure and compare implementation strategies for scaling up proven interventions. Stages range from Engagement (Stage 1) to achievement of program delivery with Competency (Stage 8). SIC data include a log of activities that operationalize the implementation process necessary to move toward successful program start-up and sustainment, and their completion dates. Two scores are calculated for each SIC stage. The Proportion score calculates the proportion of key activities completed within a stage. The Duration score is calculated by date of entry through date of final activity completed. The Duration Score can account for activities not completed sequentially and also for being in multiple stages at a given time. A third Final Stage score indicates the final stage achieved in the implementation process (Stage 1-8).
Cost of implementation | Monthly ; Months 1 to 46
  Cost of Implementing New Strategies (COINS). Calculations of fees, expenses, and person hours necessary to complete each implementation stage.
Fidelity | Months 7,14,24,34,46
  NIATx Fidelity. The NIATx Fidelity Scale is a 19-item observational measure of adherence to the NIATx model, rating activities on a 5-point scale from 1-No evidence to 5-Extensive evidence. Scoring reflects information obtained from IF and EF perspectives using a composite of interviews, review of walk-through results, change project forms, EF or IF notes and sustainability plans.
Implementation climate | Months 1,7,14,24,34,46
  Implementation Climate Scale (ICS). Assesses the extent to which an organization prioritizes and values the implementation of an evidence based practice. Six subscales and 18 items scored on a 5-point scale from 0 - not at all, to 4 - very great extent
Implementation Leadership | Months 1,7,14,24,34,46
  Implementation Leadership Scale (ILS). Assesses a leader's support for implementation of an evidence based practice. Four subscales and 12 items scored on a 5-point scale from 0 - not at all, to 4 - very great extent

CONTACTS AND LOCATIONS:
Overall Officials: Mark McGovern, PhD, Principal Investigator — Stanford University; James H Ford II, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Washington State Healthcare Authority, Olympia, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaros S, Magid MA, Cheng H, Gassman M, Garneau HC, Ford Ii JH, McGovern M. A mixed methods analysis of clinics' perspectives on community factors influencing access to medications for opioid use disorder. Addict Sci Clin Pract. 2026 Jan 8;21(1):10. doi: 10.1186/s13722-025-00643-1. PMID 41508111
- [Derived] Cheng H, Abdel Magid M, McGovern MP, Ford JH 2nd, Manja V, Chokron Garneau H, Wagner TH. A pragmatic approach to estimating the cost to deliver and participate in implementation strategies. Implement Sci. 2025 Oct 17;20(1):44. doi: 10.1186/s13012-025-01459-y. PMID 41107954
- [Derived] Ford JH 2nd, Cheng H, Gassman M, Fontaine H, Garneau HC, Keith R, Michael E, McGovern MP. Stepped implementation-to-target: a study protocol of an adaptive trial to expand access to addiction medications. Implement Sci. 2022 Sep 29;17(1):64. doi: 10.1186/s13012-022-01239-y. PMID 36175963